CLINICAL TRIAL: NCT05998486
Title: Detecting the Rest Tremor Associated With Parkinson's Disease Using Analysis of the Muscle Contractions Rhythmicity
Acronym: TREMORHYTHM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Emilie Hutin, Co-director of laboratory, Henri Mondor University Hospital
Other Study IDs: ARM-Tremor
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Parkinson; Cerebellar Tumor; Rest Tremor; Diagnoses Disease; Movement; Abnormal, Involuntary
MeSH Terms: conditions — Cerebellar Neoplasms; Tremor; Antisocial Personality Disorder | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tremor of rest: Patient with a diagnosis of Parkinson's disease and who performed surface EMG recordings of wrist flexor-pronators and extensor-supinators analysis in Laboratories
  Interventions: Diagnostic Test: EMG in wrist flexor-pronators and extensor-supinators
- Cerebellar tremor: Patient with a diagnosis of cerebellar tremor and who performed surface EMG recordings of wrist flexor-pronators and extensor-supinators analysis in Laboratories
  Interventions: Diagnostic Test: EMG in wrist flexor-pronators and extensor-supinators

INTERVENTIONS:
Diagnostic Test: EMG in wrist flexor-pronators and extensor-supinators — The subject is asked to perform a series of tasks: resting posture, symmetrical posture arms forward, unilateral distal movement. Each task lasts 10 seconds.

SUMMARY:
Resting tremors associated with Parkinson's disease (PD) remains difficult to quantify and track during disease progression. This study propose to explore the rhythmicity of distal muscle contractions in the upper limb to characterize resting tremor and discriminate it from cerebellar tremor (CT) based on the frequency spectrum of the EMG signal.

DETAILED DESCRIPTION:
This retrospective study analyzed surface EMG recordings of wrist flexor-pronators and extensor-supinators from patients with PD or CT bilaterally in five 10-second conditions: rest with contralateral motor distraction, symmetrical arms extended forward posture with hands pronated, semi-pronation, supination, and elbows flexed with hands pronated. The rhythmicity index (RI) is calculated from the ratio of the area of the maximum power peak to the total area of the spectrum between 1.5-12Hz.

ELIGIBILITY:
Inclusion Criteria:

* patient who performed surface EMG recordings of wrist flexor-pronators and extensor-supinators in Laboratories;
* diagnosis of Parkinson's disease or cerebellar tremor.

Exclusion Criteria:

* Botulinium toxin injection in upper limb during a delay of 3 months before surface EMG recordings;
* Levodopa drugs administrated during a delay of 12 hours before surface EMG recordings;
* Tremor-favour drugs administrated during a delay of 30 days before surface EMG recordings;
* Presence of an other neurologic disease or of any disease associated with motor disorders in upper limb.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease or cerebellar tremor diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
rhythmicity index | 10 seconds
  The rhythmicity index (RI) is calculated from the ratio of the area of the maximum power peak to the total area of the spectrum between 1.5-12Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Hutin, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Laboratoire Analyse et Restauration du Mouvement, Créteil, France

IPD SHARING:
Plan to Share IPD: No